CLINICAL TRIAL: NCT07052669
Title: Hypofractionated Chemoradiotherapy Followed by Consolidative Immunotherapy Versus Conventional Fractionated Chemoradiotherapy Followed by Consolidative Immunotherapy in Locally Advanced Non-small Cell Lung Cancer: A Randomized, Phase III Controlled Study
Brief Title: Hypofractionated Versus Conventional Chemoradiotherapy Followed by Consolidative Immunotherapy in Locally Advanced NSCLC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-10134
Record Dates: First submitted 2025-06-30; First posted 2025-07-06 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced Non-Small Cell Lung Cancer
Keywords: Hypofractionated radiotherapy; Conventionally fractionated radiotherapy; Concurrent Chemoradiotherapy; Consolidative immunotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypofractionated CCRT (Experimental): All patients will receive hypofractionated concurrent chemoradiotherapy, followed by consolidative immunotherapy for a maximum duration of 12 months.
  Interventions: Radiation: Hypofractionated Radiation Therapy; Drug: Concurrent Chemotherapy; Drug: Consolidative immunotherapy
- Conventional fractionated CCRT (Active Comparator): All patients will receive conventional fractionated concurrent chemoradiotherapy, followed by consolidative immunotherapy for a maximum duration of 12 months.
  Interventions: Radiation: Conventionally Fractionated Radiation Therapy; Drug: concurrent chemotherapy; Drug: Consolidative immunotherapy

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — All patients will receive split-course hypofractionated radiotherapy. First course of radiotherapy: Total dose of 4000 cGy in 10 daily fractions (400 cGy per fraction) or 3000 cGy in 6 daily fractions (500 cGy per fraction). Three weeks after the completion of the first course of hypofractionated radiotherapy, tumor response and toxicity will be evaluated. For patients who achieve a partial response and without grade 2 or higher respiratory toxicity, a second course of radiotherapy will be planned for the residue disease at a total dose of 2000 ~2400 cGy in 5~6 fractions (400 cGy per fraction). The interval between the two courses of radiotherapy will be 28 days.
  Arms: Hypofractionated CCRT
Radiation: Conventionally Fractionated Radiation Therapy — Patients in this group will receive a total dose of 6000- 6400 cGy in 30- 32 fractions, with 200 cGy per fraction.
  Arms: Conventional fractionated CCRT
Drug: Concurrent Chemotherapy — Paclitaxel plus platinum-based chemotherapy.
  Arms: Hypofractionated CCRT
Drug: concurrent chemotherapy — Paclitaxel plus platinum-based chemotherapy or pemetrexed plus platinum-based chemotherapy.
  Arms: Conventional fractionated CCRT
Drug: Consolidative immunotherapy — Following the completion of chemoradiotherapy, PD-1/PD-L1 immune checkpoint inhibitor consolidation therapy will be administered for up to 12 months.

SUMMARY:
Consolidative immunotherapy following concurrent chemoradiotherapy, based on the PACIFIC trial, has become the standard treatment for locally advanced non-small cell lung cancer (LANSCLC). Radiotherapy strategies for maximizing efficacy and local control require further investigation. This phase III, randomized controlled clinical trial is to investigate the efficacy and safety of hypofractionated chemoradiotherapy followed by consolidative immunotherapy versus conventional fractionated chemoradiotherapy followed by consolidative immunotherapy in LANSCLC patients.

DETAILED DESCRIPTION:
This phase III, randomized controlled trial aims to investigate the efficacy and safety of hypofractionated chemoradiotherapy followed by consolidative immunotherapy versus conventional fractionated chemoradiotherapy followed by consolidative immunotherapy in LANSCLC patients. Patients will be randomized in a 2:1 ratio to the following two groups: (1) Study group: Patients in this group will undergo hypofractionated chemoradiotherapy, followed by consolidative immunotherapy for a maximum duration of 12 months. (2) Control group: Patients in this group will receive conventional fractionated chemoradiotherapy followed by consolidative immunotherapy for a maximum duration of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed and Dated Informed Consent: Written informed consent must be provided prior to any study procedures, with the consent form signed and dated by the participant.
* Age Range: Male or female patients aged 18 to 75 years.
* Diagnosis: Patients must have locally advanced, unresectable (stage III) non-small cell lung cancer (NSCLC), with histological or cytological confirmation of the diagnosis.
* Previous Treatment: Treatment-naïve or previously treated with induction chemotherapy ± immunotherapy.
* Tumor Sample Requirement: Tumor tissue samples must be provided, and they should be sufficient for analysis. The samples must be unstained and archived.
* Driver gene testing: EGFR wild-type, ALK rearrangement-negative.
* Life Expectancy: Patients must have an expected survival of at least 12 weeks.
* Performance Status (PS): The patient's WHO Performance Status (PS) must be 0 or 1.
* Pregnancy Testing: Postmenopausal women, or women who have had a negative urine or serum pregnancy test within 14 days before the study medication (HCG sensitivity ≥ 25 IU/L or equivalent).
* Breastfeeding: Women must not be breastfeeding.
* Women of childbearing potential (WOCBP) must agree to use contraception during the study treatment period and for 5 months after the last dose of the investigational drug (i.e., 30 days [ovulation cycle] + approximately 5 half-lives of the study drug).
* Men who have sexual relations with WOCBP must agree to use contraception during the study treatment period and for 7 months after the last dose of the investigational drug (i.e., 90 days [sperm renewal cycle] + approximately 5 half-lives of the study drug).
* Males with no sperm production are exempt from contraception requirements. WOCBP who are not sexually active are exempt from contraception but must still undergo pregnancy testing as outlined above.
* Organ and Bone Marrow Function: The following laboratory parameters must be met:

Forced expiratory volume in 1 second (FEV1) ≥ 800 mL Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L Platelets ≥ 100 × 10⁹/L Hemoglobin ≥ 9.0 g/dL Calculated creatinine clearance using the Cockcroft-Gault formula ≥ 50 mL/min Serum bilirubin ≤ 1.5 × upper limit of normal (ULN) AST and ALT ≤ 2.5 × ULN

Exclusion Criteria:

* Patients meeting any of the following criteria should not be enrolled in the study:
* Concurrent participation in another clinical trial, except for observational (non-interventional) studies.
* Histological subtype of mixed small-cell and non-small-cell lung cancer. Use of immunosuppressive drugs within 28 days before treatment, except for intranasal or inhaled corticosteroids at physiological doses or systemic corticosteroids ≤10 mg/day of prednisone or equivalent.
* Major surgery within 4 weeks prior to enrollment (excluding procedures for vascular access).
* History or active autoimmune diseases within the past two years.
* Active or a history of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
* History of primary immunodeficiency.
* History of organ transplantation requiring immunosuppressive therapy.
* Average corrected QT interval (QTc) ≥470 ms calculated from three ECG cycles using the Bazett formula.
* Uncontrolled comorbidities, including but not limited to: Persistent or active infections. Symptomatic congestive heart failure. Poorly controlled hypertension. Unstable angina. Cardiac arrhythmias. Active peptic ulcer disease or gastritis. Active bleeding disorders. Hepatitis C or HIV infection. HBsAg-positive patients with HBV DNA >500 IU/mL. Mental or social conditions that may limit adherence to study requirements or compromise the ability to provide informed consent.
* Known history of tuberculosis.
* Receipt of a live attenuated vaccine within 30 days before study initiation or planned during the study period.
* History of another primary malignancy within the past 5 years, except for adequately treated basal or squamous cell carcinoma of the skin or in situ cervical cancer.
* Pregnancy, breastfeeding, or not using effective contraception (for men and women of reproductive potential).

Patients in the experimental group should not proceed to concurrent chemoradiotherapy if any of the following criteria are met:

* Presence of distant metastases.
* Locoregional progression making definitive concurrent chemoradiotherapy unfeasible due to normal tissue dose constraints (assessed by the radiation oncologist).
* WHO performance status score of 2-4.
* Impaired organ or bone marrow function, including:

Forced expiratory volume in 1 second (FEV1) <800 mL. Absolute neutrophil count (ANC) <1.5 × 10⁹/L. Platelets <100 × 10⁹/L. Hemoglobin <9.0 g/dL. Creatinine clearance (Cockcroft-Gault formula) <50 mL/min. Serum bilirubin >1.5 × upper limit of normal (ULN). AST and ALT >2.5 × ULN.

- Patient withdrawal from the study.

Patients should not proceed to consolidation immunotherapy if any of the following criteria are met:

* Disease progression during concurrent chemoradiotherapy.
* Use of immunosuppressive drugs within 28 days before the first dose of tislelizumab, except for physiological doses of intranasal or inhaled corticosteroids or systemic corticosteroids ≤10 mg/day of prednisone or equivalent. Use of corticosteroids to manage chemoradiotherapy-related toxicity is permitted.
* Persistent unresolved CTCAE grade >2 toxicities from prior chemoradiotherapy.
* Grade ≥2 pneumonitis resulting from prior chemoradiotherapy.
* Any prior grade ≥3 immune-related adverse event (irAE) or unresolved irAE > grade 1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Median Progression-Free Survival | 2 years
  PFS measures the time from the start of treatment until the disease progresses or the patient dies from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 1-2 months after treatment
  ORR refers to the proportion of patients who experience complete response (CR) and partial response (PR)
Overall survival (OS) | 2 years
  OS is the time from the start of treatment until death from any cause.
Failure patterns | 2 years
  Failure patterns describe the pattern of disease progression or treatment failure, such as local recurrence or distant metastases.
Safety: Adverse Events | 1 years after treatment
  Safety endpoints assess the frequency and severity of treatment-related adverse events. Adverse events are graded on a scale from 1 to 5 according to CTCAE 5.0.
Quality of life assessed by Quality of Life Core 30 | 1 years after treatment
  Patient-reported quality of life measured by European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). Higher scores on functioning scales indicate better functioning, while higher scores on symptom scales indicate more severe symptoms.
Quality of life assessed by Quality of Life LC13 | 1 years after treatment
  Patient-reported quality of life measured by European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-LC13). Higher scores on functioning scales indicate better functioning, while higher scores on symptom scales indicate more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Professor, Principal Investigator — Sun yat-sen universtiy cancer center
Locations (3):
- China (3):
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - Sun yat-sen University Cancer Center, Guangzhou, Guangdong

REFERENCES:
- [Background] Zhou R, Liu F, Zhang H, Wang D, Zhang P, Zheng S, Liu Y, Chen L, Guo J, Zou Y, Rong YM, Liu H, Qiu B. Fraction Dose Escalation of Hypofractionated Radiotherapy with Concurrent Chemotherapy and Subsequent Consolidation Immunotherapy in Locally Advanced Non-Small Cell Lung Cancer: A Phase I Study. Clin Cancer Res. 2024 Jul 1;30(13):2719-2728. doi: 10.1158/1078-0432.CCR-23-3600. PMID 38652815
- [Background] Filatenkov A, Baker J, Mueller AM, Kenkel J, Ahn GO, Dutt S, Zhang N, Kohrt H, Jensen K, Dejbakhsh-Jones S, Shizuru JA, Negrin RN, Engleman EG, Strober S. Ablative Tumor Radiation Can Change the Tumor Immune Cell Microenvironment to Induce Durable Complete Remissions. Clin Cancer Res. 2015 Aug 15;21(16):3727-39. doi: 10.1158/1078-0432.CCR-14-2824. Epub 2015 Apr 13. PMID 25869387
- [Background] Lee Y, Auh SL, Wang Y, Burnette B, Wang Y, Meng Y, Beckett M, Sharma R, Chin R, Tu T, Weichselbaum RR, Fu YX. Therapeutic effects of ablative radiation on local tumor require CD8+ T cells: changing strategies for cancer treatment. Blood. 2009 Jul 16;114(3):589-95. doi: 10.1182/blood-2009-02-206870. Epub 2009 Apr 6. PMID 19349616
- [Background] Tang C, Liao Z, Gomez D, Levy L, Zhuang Y, Gebremichael RA, Hong DS, Komaki R, Welsh JW. Lymphopenia association with gross tumor volume and lung V5 and its effects on non-small cell lung cancer patient outcomes. Int J Radiat Oncol Biol Phys. 2014 Aug 1;89(5):1084-1091. doi: 10.1016/j.ijrobp.2014.04.025. Epub 2014 Jul 8. PMID 25035212
- [Background] Wild AT, Herman JM, Dholakia AS, Moningi S, Lu Y, Rosati LM, Hacker-Prietz A, Assadi RK, Saeed AM, Pawlik TM, Jaffee EM, Laheru DA, Tran PT, Weiss MJ, Wolfgang CL, Ford E, Grossman SA, Ye X, Ellsworth SG. Lymphocyte-Sparing Effect of Stereotactic Body Radiation Therapy in Patients With Unresectable Pancreatic Cancer. Int J Radiat Oncol Biol Phys. 2016 Mar 1;94(3):571-9. doi: 10.1016/j.ijrobp.2015.11.026. Epub 2015 Dec 1. PMID 26867885
- [Background] Zhou R, Qiu B, Xiong M, Liu Y, Peng K, Luo Y, Wang D, Liu F, Chen N, Guo J, Zhang J, Huang X, Rong Y, Liu H. Hypofractionated Radiotherapy followed by Hypofractionated Boost with weekly concurrent chemotherapy for Unresectable Stage III Non-Small Cell Lung Cancer: Results of A Prospective Phase II Study (GASTO-1049). Int J Radiat Oncol Biol Phys. 2023 Oct 1;117(2):387-399. doi: 10.1016/j.ijrobp.2023.04.021. Epub 2023 Apr 25. PMID 37100160
- [Background] Kong FM, Ten Haken RK, Schipper M, Frey KA, Hayman J, Gross M, Ramnath N, Hassan KA, Matuszak M, Ritter T, Bi N, Wang W, Orringer M, Cease KB, Lawrence TS, Kalemkerian GP. Effect of Midtreatment PET/CT-Adapted Radiation Therapy With Concurrent Chemotherapy in Patients With Locally Advanced Non-Small-Cell Lung Cancer: A Phase 2 Clinical Trial. JAMA Oncol. 2017 Oct 1;3(10):1358-1365. doi: 10.1001/jamaoncol.2017.0982. PMID 28570742
- [Background] Durm GA, Jabbour SK, Althouse SK, Liu Z, Sadiq AA, Zon RT, Jalal SI, Kloecker GH, Williamson MJ, Reckamp KL, Langdon RM, Kio EA, Gentzler RD, Adesunloye BA, Harb WA, Walling RV, Titzer ML, Hanna NH. A phase 2 trial of consolidation pembrolizumab following concurrent chemoradiation for patients with unresectable stage III non-small cell lung cancer: Hoosier Cancer Research Network LUN 14-179. Cancer. 2020 Oct 1;126(19):4353-4361. doi: 10.1002/cncr.33083. Epub 2020 Jul 22. PMID 32697352
- [Background] Spigel DR, Faivre-Finn C, Gray JE, Vicente D, Planchard D, Paz-Ares L, Vansteenkiste JF, Garassino MC, Hui R, Quantin X, Rimner A, Wu YL, Ozguroglu M, Lee KH, Kato T, de Wit M, Kurata T, Reck M, Cho BC, Senan S, Naidoo J, Mann H, Newton M, Thiyagarajah P, Antonia SJ. Five-Year Survival Outcomes From the PACIFIC Trial: Durvalumab After Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. J Clin Oncol. 2022 Apr 20;40(12):1301-1311. doi: 10.1200/JCO.21.01308. Epub 2022 Feb 2. PMID 35108059
- [Background] Gray JE, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Kurata T, Chiappori A, Lee KH, Cho BC, Planchard D, Paz-Ares L, Faivre-Finn C, Vansteenkiste JF, Spigel DR, Wadsworth C, Taboada M, Dennis PA, Ozguroglu M, Antonia SJ. Three-Year Overall Survival with Durvalumab after Chemoradiotherapy in Stage III NSCLC-Update from PACIFIC. J Thorac Oncol. 2020 Feb;15(2):288-293. doi: 10.1016/j.jtho.2019.10.002. Epub 2019 Oct 14. PMID 31622733
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881